CLINICAL TRIAL: NCT04802720
Title: A Randomized Controlled Trial of Emotion Regulation Therapy for Cancer Caregivers: A Mechanism-Targeted Approach to Addressing Caregiver Distress
Brief Title: A Study Comparing Two Types of Supportive Interventions for Caregivers of Patients With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Aarhus (Other); Columbia University (Other); University of California (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-407
Record Dates: First submitted 2021-03-01; First posted 2021-03-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cancer Patients; Family Caregivers
Keywords: Emotion Regulation Therapy; Addressing Caregiver Distress; Supportive Interventions; 20-407; Training participants
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized, controlled, repeated measures design to investigate the efficacy of Emotion Regulation Therapy for Cancer Caregivers (ERT-C) vs. Cognitive Behavioral Therapy for Cancer Caregivers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ERT-C: Emotion Regulation Therapy for Cancer Caregivers (Experimental): Emotion Regulation Therapy for Cancer Caregivers (ERT-C) is an 8-session intervention that builds upon the foundations of CBT-C and addresses earlier motivational processing components of the caregivers context while targeting earlier and later components of internal distress and resultant maladaptive behavioral coping.
  Interventions: Other: Emotion Regulation Therapy for Cancer Caregivers (ERT-C)
- CBT-C: Cognitive Behavioral Therapy for Cancer Caregivers (Experimental): Cognitive Behavioral Therapy (CBT-C) is an evidence-based psychotherapeutic approach that is grounded in the cognitive model that purports that a person's emotional, behavioral, and physiological reactions to a situation is based on their appraisal of that situation. The focus of therapy is on changing cognitions and beliefs about a situation and altering automatic behavioral responses evoked by that perception. CBT-C aims to improve emotion regulation by challenging and changing unhelpful cognitions and behaviors and improving personal coping strategies.
  Interventions: Other: Cognitive Behavioral Therapy for Cancer Caregivers (CBT-C)
- Training case group (Experimental): Will be assigned to receive ERT-C only and will not complete questionnaires.
  Interventions: Other: Emotion Regulation Therapy for Cancer Caregivers (ERT-C)

INTERVENTIONS:
Other: Cognitive Behavioral Therapy for Cancer Caregivers (CBT-C) — The sessions are outlined as follow:
  1. psychoeducation, goal-setting, and describing the rationale for CBT (Session 1);
  2. coping effectiveness training (Session 2);
  3. identifying unhelpful cognitions and dysfunctional beliefs (Session 3);
  4. challenging and restructuring unhelpful cognitions (Session 4);
  5. behavioral activation within the limitations of the caregiving context (Session 5);
  6. problem-solving (Session 6);
  7. communication strategies and assertiveness training (Session 7);
  8. consolidating gains, maintenance, and relapse prevention (Session 8).
  Arms: CBT-C: Cognitive Behavioral Therapy for Cancer Caregivers
Other: Emotion Regulation Therapy for Cancer Caregivers (ERT-C) — The sessions are outlined as follow:
  1. psychoeducation and motivation/dysregulation cue detection within caregiving contexts (Session 1);
  2. attention regulation skills training (Sessions 1-2);
  3. training in metacognitive skills (Sessions 3-4);
  4. exposure to proactive living in the face of risk and loss while applying skills (Sessions 5-7);
  5. consolidating gains, taking larger proactive steps, and relapse prevention (Session 8).
  Arms: ERT-C: Emotion Regulation Therapy for Cancer Caregivers; Training case group

SUMMARY:
The purpose of this study is to compare two types of therapy for caregivers of cancer patients: Emotion Regulation Therapy for Cancer Caregivers (ERT-C) and Cognitive Behavioral Therapy (CBT-C). The researchers want to see if ERT-C is better than, the same as, or worse than traditional CBT-C at improving caregiver distress. The researchers will look at how the two types of therapy affect caregivers' anxiety, depression, and quality of life. The researchers will also see how ERT-C and CBT-C affect hormone and stress levels in caregivers' saliva samples.

In addition, this trial will enroll cancer patients in this study to see how their caregivers' participation in ERT-C or CBT may affect the patients' quality of life, stress, and use of healthcare services.

Participants who become bereaved while on study will be given the option to withdraw or remain on study. Assessments for bereaved caregivers will not include the Caregiver Quality of Life Index-Cancer (CQOLC) or the Caregiver Reaction Assessment (CRA).

DETAILED DESCRIPTION:
CBT-C and ERT-C are each 8-session, individual, caregivers-directed interventions delivered by a trained study therapist listed on the face page and facilitated by a manualized workbook with between-session practice exercises. To accommodate caregivers and reduce compliance issues with attendance of sessions, the 8 sessions are to be completed within 8 to 16 weeks from initiation of the first session. Each session is 60 minutes in length and will be audio and video recorded for MSK participants; sessions will only be audio recorded for MGH participants. Specific modules and intervention components are described below. To accommodate as many caregivers as possible and in response to the restrictions placed on caregivers currently in the context of the COVID-19 pandemic, sessions will be offered via telepsychiatry (using WebEx , Zoom, Teams).

Training case participants will be identified and consented onto the study for training purposes only. Participants who are consented as training cases will not be randomized and will not complete any assessments. Data collected on training cases will be used for training and supervision purposes on this study only. These records will not be shown outside of the study supervisors, therapist in training, and staff.

ELIGIBILITY:
Inclusion Criteria:

Caregivers:

* As per self-report, age 18 years or older.
* As per self-report, are a caregiver to an MSK or MGH patient with any site/stage of cancer who has received any type of treatment (e.g. curative, palliative) in the past 12 months.
* Experience distress as evidenced by a score of 4 or greater on the Distress Thermometer (DT) and answer "Yes" to at least one of the follow-up questions (i.e. reporting that their distress is related to their caregiving experience, or their distress started or is related to caregiving or has gotten worse since the patient was diagnosed or began treatment. (N/A for training case participants)
* English fluent: Self-report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* As per self-report, residing in New York or New Jersey (for MSK participants), or Massachusetts (for MGH participants), or have the ability to complete sessions while complying with current telehealth regulations.

Patients:

* Age 18 years or older as per EMR.
* Patient of an eligible caregiver per self-report or the EMR.
* English speaking as per the EMR or self report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well.".

Exclusion Criteria:

Caregivers:

* As per self-report, presence of disorder that compromises comprehension of assessments or informed consent information (e.g., dementia).
* As per the judgement of the consenting professional, clinical, PI, and/or as per the medical record, severe psychopathology or cognitive impairment which is likely to interfere with the participation or completion of the protocol or their ability to provide meaningful information
* As per self-report, currently engaged in regular individual psychotherapeutic support (that the participant is unable or unwilling to put on hold for the course of treatment).
* As per self-report, a lifetime history of bipolar disorder, schizophrenia, or schizoaffective disorder.
* As per self-report, has medical condition or medication use known to confound measures of systemic inflammation (e.g., autoimmune disorder, inflammatory disease; uncontrolled thyroid disease; active infection; myocardial infarction or stroke in the last 6 months; Type I diabetes; acute hepatitis; recent vaccination for viral disease). (N/A for training case participants)
* As per self-report, is a regular smoker, defined as having more than 2 cigarettes per day on most days. (N/A for training case participants)
* As per self-report, providing care for a patient who has a caregiver is currently or formerly enrolled in this study ('formerly enrolled' is N/A for training case participants).
* As per self-report, currently enrolled in another study focused on supportive care for caregivers (MGH participants only).

Patients:

* Presence of disorder that compromises comprehension of assessments or informed consent information (e.g., dementia) as per EMR or clinician judgment.
* As per the judgement of the consenting professional, clinical, PI, and/or as per the medical record, severe psychopathology or cognitive impairment which is likely to interfere with the participation or completion of the protocol or their ability to provide meaningful information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
changes in anxiety symptoms | up to 6 months
  as assessed via the HADS Developed by Zigmond and Snaith in 1983, the HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Items of the overall severity of anxiety and depression are rated on a five-point (0-4) severity scales (ranging from 0 = no not at all, to 3 = yes definitely), for a total score ranging from 0-21 for each subscale. A higher score indicates higher distress
changes in depressive symptoms | up to 6 months
  as assessed via the HADS Developed by Zigmond and Snaith in 1983, the HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Items of the overall severity of anxiety and depression are rated on a five-point (0-4) severity scales (ranging from 0 = no not at all, to 3 = yes definitely), for a total score ranging from 0-21 for each subscale. A higher score indicates higher distress

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of California, Irvine (Data and Specimen Analysis Only), Irvine, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Hospital (Data Analysis Only), New York, New York
  - Columbia University (Data and Specimen Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04802720/ICF_000.pdf